CLINICAL TRIAL: NCT04797078
Title: Prospective Randomized Controlled Study: Free-Hand Transperineal vs. Transrectal Systematic and Image Fusion Targeted Biopsies Under Local Anesthesia Comparing Rate of Significant Cancer Detection and Complication Rates
Brief Title: US/MRI Fusion Local Anestesia TransPerineal Prostate Biopsies for Detection of Prostate Cancer
Acronym: FLAPP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Planning halted due to changes in the research group constellation.
Sponsor: Karolinska Institutet (Other)
Collaborators: Capio Sankt Görans Hospital (Other); GHP Urologi Odenplan (Unknown); Urologifocus Stockholm (Unknown)
Responsible Party: Principal Investigator, Tobias Nordström, MD PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STHLM3FLAPP
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Prostate Cancer
Keywords: transperineal biopsy; prostate cancer detection
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transrectal fusion biopsies of the prostate (Active Comparator): 1. Transrectal approach, patient in left lateral position, local anestesia 10ml lidocaine 1% at prostate base laterally and apex if indicated.
  2. MRI-ultrasound fusion-guided biopsies with 4 biopsy cores per lesion, where clinically indicated. 18G biopsy needle.
  3. Standard 12-core template for systematic biopsies. 18G biopsy needle.
  4. Antibiotic prophylaxis with 750mg ciprofloxaicin, single dose p.o.
  Interventions: Procedure: Transrectal biopsy
- Transperineal free hand fusion biopsies of the prostate (Experimental): Men randomized to the experimental arm undergoes free-hand targeted transperineal fusion biopsies as defined below.
  1. Patient is placed supine in the lithotomy-position. The perineal area is prepared with chlorhexidine 0,5ml/ml.
  2. Ropivacain 7,5mg/ml is used as an anesthetic agent. Up to 40ml's (equivalent to 300mg) can be used to anestitize the skin, caudal and cranial part of the urogenital diaphragm and periprostatic tissue.
  3. Free-hand MRI-ultrasound fusion-guided biopsies with at least 4 biopsy cores per lesion. Coaxial technique with 18G biopsy needle.
  4. 10-12 Systematic biopsies according to the modified Barzell 12-core template.
  5. No antibiotic profylaxis unless warranted by immunosuppression, previous sepsis or urinary tract infection.
  Interventions: Procedure: Transperineal biopsy

INTERVENTIONS:
Procedure: Transperineal biopsy — Transperineal free hand MRI-US fusion prostate biopsy
  Arms: Transperineal free hand fusion biopsies of the prostate
Procedure: Transrectal biopsy — Transrectal MRI-US fusion prostate biopsy
  Arms: Transrectal fusion biopsies of the prostate

SUMMARY:
We are conducting a randomised trial comparing outcomes of transperineal prostate biopsies under free-hand software assisted MRI/US fusion with transrectal biopsy guide software assisted MRI/US fusion. Primary outcome is the detection of clinically significant prostate cancer. Secondary outcomes is rate of complications including infection and sepsis, as well as feasibility and patient tolerability.

DETAILED DESCRIPTION:
Prostate cancer is a leading cause of cancer death among men in the Western world. Early detection of prostate cancer has been shown to decrease mortality. When a test for prostate cancer yields an elevated risk of prostate cancer, tissue sampling from the prostate is warranted. The common practice is to acquire these biopsies has been via transrectal biopsies under ultrasound guidance (TRUL-biopsies). A low estimate of the risk of hospital-requiring infection is 5%, yielding unnecessary and costly sepsis cases.

In addition to suffering and loss of production, as well as healthcare costs, in a material from Taiwan, the mortality risk of biopsy-induced sepsis has been estimated at 0.13%. In a publication from Norway, it is estimated that infection complications from tissue sampling of the prostate cause 10 deaths per year (population 5 million).

Previous international studies show that the risk of infection with bacteria from the gut can be completely eliminated by taking the tissue samples through the skin of the perineum, transperineal biopsies (TPb), with guidance from transrectal ultrasound. This method is well established for systematic biopsies and has been proven safe in large series.

Studies have showed how multiparametric magnetic-resonance imaging (mpMRI) of the prostate accurately can identify lesions harboring clinically significant prostate cancer (csPC, defined as ISUP Gleason Group (GG) ≥ 2)3. Prostate MRI reading and reporting according to the PI-RADS protocol is widely accepted and recommended.

The image material from the MRI can be used to produce maps of the prostate used for tissue sampling of suspected areas. This is referred to as MRI/ultrasound fusion biopsy, or targeted biopsies (TBx). Regions of interest are marked as Lesions. Several studies have shown improved cancer detection using MRI and fusion targeted biopsies in clinical-practice cohorts 5,6 78 MRI/ultrasound fusion biopsies can be performed in a variety of ways, where software assisted transrectal biopsies has gained the most attention during the last few years, earning to development of equipment more readily available to the urologist as well as a rise in the quantity and quality of prostate MRI's.

The combination of transperineal prostate biopsies and targeted biopsies can be done with a rigid system of stepper and brachy-grid guiding. Recently, several systems for free-hand transperineal biopsies have been introduced, but data and recommendations on biopsy strategies and accuracy is lacking. The detection rates of cancer has not been evaluated in In comparison with transrectal prostate biopsy, transperineal prostate biopsy has the advantage of better sampling from the anterior area of the prostate, an area that is technically more challenging to sample with the transrectal approach. Other advantages of the transperineal route is believed to be the low risk of infection, and no risk ofrectal bleeding. The main challenge associated with the transperineal method is patient discomfort and pain management.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent to participate
* Be aged 18 years and over
* An understanding of the Swedish language sufficient to understand written and verbal information about the trial and consent process
* Be suited and fit for either procedure (transrectal/transperineal)
* Be suitable for a prostate biopsy and clinically due to have a biopsy for diagnostic purpose (following indications for biopsy)

  * Biopsy naïve
  * Men on active surveillance (AS)
  * Rebiopsy
* Be willing and able to comply with scheduled visits and completion of study questionnaires

Exclusion Criteria:

* Severe illness such as metastatic cancers, sever cardio-vascular disease or dementia
* Men with contraindication for a prostate biopsy
* Men without suspect lesions on MRI
* Previous TURP or other BPH treatment (HoLEP, PostaLUND, water-vaporization) is permitted, but men who have had HIFU, cryo, IRE (irreversible electroporation), photodynamic, or microwave therapy to the prostate will not be included.
* Previous treatment with BCG for bladder cancer
* Men who are unable to undergo transrectal ultrasonography
* Men who have had previous radiation therapy to the pelvis
* Men not tolerating ciprofloxacin
* Unable to lie down with legs in a stirrup for at least 45 minutes, as assessed by a clinician

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Rate of prostate cancer detection | Data available at completed inclusion
  Detection of clinically significant prostate cancer (defined as any ISUP >2). Per PIRADS grade group.

SECONDARY OUTCOMES:
Rate of urinary tract infection and sepsis | Data available at completed inclusion + 30 days
  Rate of infectious complications (defined as treatment with antibiotics) within 30 days after intervention. Stratified on infections requiring hospitalization.
Individual complications requiring hospital admission. | Data available at completed inclusion + 30 days
  Any complication after intervention requiring hotspital admission within 30 days

OTHER OUTCOMES:
Patient tolerability | Data available at completed inclusion + 30 days
  * Pain level assessed by visual analogue scale (VAS)
  * Most painful part of procedure
  * Assessed immediately following procedure, and at 30 days
Outcomes after radical prostatectomy | 1 yr after study inclusion closes
  Rate of radical surgery and functional outcomes after radical prostatectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Nordström, PhD, Principal Investigator — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Culp MB, Soerjomataram I, Efstathiou JA, Bray F, Jemal A. Recent Global Patterns in Prostate Cancer Incidence and Mortality Rates. Eur Urol. 2020 Jan;77(1):38-52. doi: 10.1016/j.eururo.2019.08.005. Epub 2019 Sep 5. PMID 31493960
- [Background] Chiu PK, Alberts AR, Venderbos LDF, Bangma CH, Roobol MJ. Additional benefit of using a risk-based selection for prostate biopsy: an analysis of biopsy complications in the Rotterdam section of the European Randomized Study of Screening for Prostate Cancer. BJU Int. 2017 Sep;120(3):394-400. doi: 10.1111/bju.13913. Epub 2017 Jun 5. PMID 28498624
- [Background] Turkbey B, Rosenkrantz AB, Haider MA, Padhani AR, Villeirs G, Macura KJ, Tempany CM, Choyke PL, Cornud F, Margolis DJ, Thoeny HC, Verma S, Barentsz J, Weinreb JC. Prostate Imaging Reporting and Data System Version 2.1: 2019 Update of Prostate Imaging Reporting and Data System Version 2. Eur Urol. 2019 Sep;76(3):340-351. doi: 10.1016/j.eururo.2019.02.033. Epub 2019 Mar 18. PMID 30898406
- [Background] Alberts AR, Roobol MJ, Verbeek JFM, Schoots IG, Chiu PK, Osses DF, Tijsterman JD, Beerlage HP, Mannaerts CK, Schimmoller L, Albers P, Arsov C. Prediction of High-grade Prostate Cancer Following Multiparametric Magnetic Resonance Imaging: Improving the Rotterdam European Randomized Study of Screening for Prostate Cancer Risk Calculators. Eur Urol. 2019 Feb;75(2):310-318. doi: 10.1016/j.eururo.2018.07.031. Epub 2018 Aug 3. PMID 30082150
- [Background] Drost FH, Osses DF, Nieboer D, Steyerberg EW, Bangma CH, Roobol MJ, Schoots IG. Prostate MRI, with or without MRI-targeted biopsy, and systematic biopsy for detecting prostate cancer. Cochrane Database Syst Rev. 2019 Apr 25;4(4):CD012663. doi: 10.1002/14651858.CD012663.pub2. PMID 31022301
- [Background] Ahmed HU, El-Shater Bosaily A, Brown LC, Gabe R, Kaplan R, Parmar MK, Collaco-Moraes Y, Ward K, Hindley RG, Freeman A, Kirkham AP, Oldroyd R, Parker C, Emberton M; PROMIS study group. Diagnostic accuracy of multi-parametric MRI and TRUS biopsy in prostate cancer (PROMIS): a paired validating confirmatory study. Lancet. 2017 Feb 25;389(10071):815-822. doi: 10.1016/S0140-6736(16)32401-1. Epub 2017 Jan 20. PMID 28110982
- [Background] Kasivisvanathan V, Rannikko AS, Borghi M, Panebianco V, Mynderse LA, Vaarala MH, Briganti A, Budaus L, Hellawell G, Hindley RG, Roobol MJ, Eggener S, Ghei M, Villers A, Bladou F, Villeirs GM, Virdi J, Boxler S, Robert G, Singh PB, Venderink W, Hadaschik BA, Ruffion A, Hu JC, Margolis D, Crouzet S, Klotz L, Taneja SS, Pinto P, Gill I, Allen C, Giganti F, Freeman A, Morris S, Punwani S, Williams NR, Brew-Graves C, Deeks J, Takwoingi Y, Emberton M, Moore CM; PRECISION Study Group Collaborators. MRI-Targeted or Standard Biopsy for Prostate-Cancer Diagnosis. N Engl J Med. 2018 May 10;378(19):1767-1777. doi: 10.1056/NEJMoa1801993. Epub 2018 Mar 18. PMID 29552975
- [Background] Loeb S, Vellekoop A, Ahmed HU, Catto J, Emberton M, Nam R, Rosario DJ, Scattoni V, Lotan Y. Systematic review of complications of prostate biopsy. Eur Urol. 2013 Dec;64(6):876-92. doi: 10.1016/j.eururo.2013.05.049. Epub 2013 Jun 4. PMID 23787356
- [Background] Grummet J, Gorin MA, Popert R, O'Brien T, Lamb AD, Hadaschik B, Radtke JP, Wagenlehner F, Baco E, Moore CM, Emberton M, George AK, Davis JW, Szabo RJ, Buckley R, Loblaw A, Allaway M, Kastner C, Briers E, Royce PL, Frydenberg M, Murphy DG, Woo HH. "TREXIT 2020": why the time to abandon transrectal prostate biopsy starts now. Prostate Cancer Prostatic Dis. 2020 Mar;23(1):62-65. doi: 10.1038/s41391-020-0204-8. Epub 2020 Jan 13. No abstract available. PMID 31932659
- [Background] Kum F, Elhage O, Maliyil J, Wong K, Faure Walker N, Kulkarni M, Namdarian B, Challacombe B, Cathcart P, Popert R. Initial outcomes of local anaesthetic freehand transperineal prostate biopsies in the outpatient setting. BJU Int. 2020 Feb;125(2):244-252. doi: 10.1111/bju.14620. Epub 2019 Dec 3. PMID 30431694
- [Background] Kuru TH, Wadhwa K, Chang RT, Echeverria LM, Roethke M, Polson A, Rottenberg G, Koo B, Lawrence EM, Seidenader J, Gnanapragasam V, Axell R, Roth W, Warren A, Doble A, Muir G, Popert R, Schlemmer HP, Hadaschik BA, Kastner C. Definitions of terms, processes and a minimum dataset for transperineal prostate biopsies: a standardization approach of the Ginsburg Study Group for Enhanced Prostate Diagnostics. BJU Int. 2013 Sep;112(5):568-77. doi: 10.1111/bju.12132. Epub 2013 Jun 17. PMID 23773772
- [Background] Chiu PK, Lo KL, Teoh JY, Ma SF, Leung CH, Wong HF, Li KM, Sae-Lo K, Kwok SW, Li SY, Yee CH, Hou SM, Ng CF. Sectoral cancer detection and tolerability of freehand transperineal prostate biopsy under local anaesthesia. Prostate Cancer Prostatic Dis. 2021 Jun;24(2):431-438. doi: 10.1038/s41391-020-00293-1. Epub 2020 Sep 30. PMID 32999465
- [Background] Epstein JI, Egevad L, Amin MB, Delahunt B, Srigley JR, Humphrey PA; Grading Committee. The 2014 International Society of Urological Pathology (ISUP) Consensus Conference on Gleason Grading of Prostatic Carcinoma: Definition of Grading Patterns and Proposal for a New Grading System. Am J Surg Pathol. 2016 Feb;40(2):244-52. doi: 10.1097/PAS.0000000000000530. PMID 26492179